CLINICAL TRIAL: NCT00741793
Title: BioTRAC (BIOLOGIC TREATMENT REGISTRY ACROSS CANADA)
Brief Title: Biologic Treatment Registry Across Canada
Acronym: BioTRAC
Status: Completed | Type: Observational
Sponsor: Janssen Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR100762; P02843 (Other: Janssen Inc.)
Record Dates: First submitted 2008-08-22; First posted 2008-08-26 (Estimated); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Arthritis, Rheumatoid; Spondyloarthritis, Axial; Arthritis, Psoriatic
Keywords: Rheumatoid arthritis; psoriatic arthritis; axial spondyloarthritis; Remicade®; Simponi®; Simponi® I.V; Stelara®; Registry; BioTRAC
MeSH Terms: conditions — Arthritis, Rheumatoid; Axial Spondyloarthritis; Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

SUMMARY:
This registry is a multi-center, prospective, longitudinal, observational program that will gather and analyse data on participants treated with infliximab, golimumab, golimumab Intravenous (I.V) or ustekinumab. Treatment will be prescribed by the physician according to actual clinical practice or standard of care for Rheumatoid Arthritis (RA), Axial Spondyloarthritis (AxSpA) , Psoriatic Arthritis (PsA); there will be no randomized assignments to treatment. At baseline and approximately every 6 months thereafter, information will be collected to assess safety, clinical outcomes, quality of life, comorbidities, pharmacoeconomics and treatment regimens among cohorts of participants receiving infliximab, golimumab, golimumab I.V or ustekinumab for the treatment of RA, AxSpA and PsA.

DETAILED DESCRIPTION:
Participants will be selected for this registry using a non-probability sampling method.

ELIGIBILITY:
Inclusion Criteria:

* Participant is starting infliximab, golimumab, golimumab Intravenous (I.V) or ustekinumab at the time of enrollment and is biologic naive or has been treated with only one prior biologic (including infliximab, golimumab, golimumab I.V or ustekinumab) prior to enrollment
* Participant has signed the approved informed consent form
* Participant is diagnosed with RA, AxSpA or PsA and is eligible for treatment with infliximab, golimumab, golimumab I.V or ustekinumab in accordance with routine clinical care and the Canadian Product Monograph.

Exclusion Criteria:

- Participant was treated with two or more biologics, for any period of time before enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with RA, AxSpA, or PsA will be selected primarily from community centers and some academic centers.
Sampling Method: Non-Probability Sample
Enrollment: 2821 (Actual)
Dates: Start 2002-02-12 (Actual); Primary Completion 2018-06-27 (Actual); Study Completion 2018-06-29 (Actual)

PRIMARY OUTCOMES:
Disease Status of Canadian Participants With Rheumatic Disease Treated With Infliximab | Up to 4 years
  Physician will rate arthritis activity using Visual Analog Scale (VAS) ranging from 0 to 100; higher scores indicated greater affectation due to disease activity.
Disease Status of Canadian Participants With Rheumatic Disease Treated With Golimumab | Up to 4 years
  Physician will rate arthritis activity using VAS ranging from 0 to 100; higher scores indicated greater affectation due to disease activity.
Disease Status of Canadian Participants With Rheumatic Disease Treated With Golimumab Intravenous (I.V) | Up to 4 years
  Physician will rate arthritis activity using VAS ranging from 0 to 100; higher scores indicated greater affectation due to disease activity.
Disease Status of Canadian Participants With Rheumatic Disease Treated With Ustekinumab | Up to 4 years
  Physician will rate arthritis activity using VAS ranging from 0 to 100; higher scores indicated greater affectation due to disease activity.

SECONDARY OUTCOMES:
The Number of Participants With Adverse Events | Up to 4 years
Expanded Information and Support for Healthcare Providers and Hospitals About the Appropriate use of Infliximab | Up to 4 years
  Provides expanded data to health care providers and hospitals to estimate and support appropriate use of Infliximab.
Expanded Information and Support for Healthcare Providers and Hospitals About the Appropriate use of Golimumab | Up to 4 years
  Provides expanded data to health care providers and hospitals to estimate and support appropriate use of Golimumab.
Expanded Information and Support for Healthcare Providers and Hospitals About the Appropriate use of Golimumab I.V | Up to 4 years
  Provides expanded data to health care providers and hospitals to estimate and support appropriate use of Golimumab I.V.
Expanded Information and Support for Healthcare Providers and Hospitals About the Appropriate use of Ustekinumab | Up to 4 years
  Provides expanded data to health care providers and hospitals to estimate and support appropriate use of Ustekinumab.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Inc. Clinical Trial, Study Director — Janssen Inc.
Locations (1):
- Montreal, Quebec, Canada

REFERENCES:
- [Derived] Arendse R, Rahman P, Baer P, Haaland D, Bessette L, Sholter D, Rachich M, Rampakakis E, Marrache AM, Lehman AJ, Asin-Milan O. Safety of Golimumab in Patients with Rheumatoid Arthritis, Psoriatic Arthritis, and Axial Spondyloarthritis: Results from a Real-World Canadian Setting. Rheumatol Ther. 2025 Dec;12(6):1043-1055. doi: 10.1007/s40744-025-00788-0. Epub 2025 Sep 19. PMID 40971024
- [Derived] Bessette L, Rahman P, Kelsall J, Purvis J, Rampakakis E, Lehman AJ, Rachich M, Nantel F, Asin-Milan O, Marrache AM. Real-World Incidence and Determinants of Infection in Patients With Rheumatoid Arthritis Treated With Golimumab After a Median Follow-Up Time of 27 Months. J Rheumatol. 2023 Sep;50(9):1121-1126. doi: 10.3899/jrheum.2022-1283. Epub 2023 Jun 1. PMID 37263649
- [Derived] Rahman P, Starr M, Haaland D, Bessette L, Teo M, Rampakakis E, Lehman AJ, Nantel F. Long-term effectiveness and safety of infliximab and golimumab in ankylosing spondylitis patients from a Canadian prospective observational registry. BMC Rheumatol. 2020 Nov 15;4(1):56. doi: 10.1186/s41927-020-00158-z. PMID 33292797
- [Derived] Rahman P, Baer P, Keystone E, Choquette D, Thorne C, Haraoui B, Chow A, Faraawi R, Olszynski W, Kelsall J, Rampakakis E, Lehman AJ, Nantel F. Long-term effectiveness and safety of infliximab, golimumab and golimumab-IV in rheumatoid arthritis patients from a Canadian prospective observational registry. BMC Rheumatol. 2020 Sep 19;4:46. doi: 10.1186/s41927-020-00145-4. eCollection 2020. PMID 32968710
- [Derived] Rahman P, Arendse R, Khraishi M, Sholter D, Sheriff M, Rampakakis E, Lehman AJ, Nantel F. Long-term effectiveness and safety of infliximab, golimumab and ustekinumab in patients with psoriatic arthritis from a Canadian prospective observational registry. BMJ Open. 2020 Aug 13;10(8):e036245. doi: 10.1136/bmjopen-2019-036245. PMID 32792436
- [Derived] Rahman P, Zummer M, Bessette L, Baer P, Haraoui B, Chow A, Kelsall J, Kapur S, Rampakakis E, Psaradellis E, Lehman AJ, Nantel F, Osborne B, Tkaczyk C. Real-world validation of the minimal disease activity index in psoriatic arthritis: an analysis from a prospective, observational, biological treatment registry. BMJ Open. 2017 Aug 30;7(8):e016619. doi: 10.1136/bmjopen-2017-016619. PMID 28855200
- [Derived] Rahman P, Choquette D, Bensen WG, Khraishi M, Chow A, Zummer M, Shaikh S, Sheriff M, Dixit S, Sholter D, Psaradellis E, Sampalis JS, Letourneau V, Lehman AJ, Nantel F, Rampakakis E, Otawa S, Shawi M. Biologic Treatment Registry Across Canada (BioTRAC): a multicentre, prospective, observational study of patients treated with infliximab for ankylosing spondylitis. BMJ Open. 2016 Apr 5;6(4):e009661. doi: 10.1136/bmjopen-2015-009661. PMID 27048632
- [Derived] Haraoui B, Jovaisas A, Bensen WG, Faraawi R, Kelsall J, Dixit S, Rodrigues J, Sheriff M, Rampakakis E, Sampalis JS, Lehman AJ, Otawa S, Nantel F, Shawi M. Use of corticosteroids in patients with rheumatoid arthritis treated with infliximab: treatment implications based on a real-world Canadian population. RMD Open. 2015 Apr 29;1(1):e000078. doi: 10.1136/rmdopen-2015-000078. eCollection 2015. PMID 26509071